CLINICAL TRIAL: NCT00056485
Title: Behavioral Intervention for Depression in Nursing Homes
Brief Title: Treatment of Depression in Nursing Homes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Louisville (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Suzanne Meeks, Professor, University of Louisville
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: R21MH063073 (NIH); R21MH063073 (NIH)
Record Dates: First submitted 2003-03-14; First posted 2003-03-17 (Estimated); Last update posted 2017-04-13 (Actual); Status verified 2017-04

CONDITIONS: Depression
Keywords: Nursing homes; Aging
MeSH Terms: conditions — Depression

STUDY DESIGN:
Intervention Model Description: This was a pilot feasibility study; the first part was a single group; the second part was a two-group randomized design.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Behavioral: Pleasant Events-Based Behavioral Intervention

SUMMARY:
This study will implement a treatment for depression in a nursing home setting.

DETAILED DESCRIPTION:
Depression in long-term care facilities is a significant public health issue. Up to 50% of nursing home residents are affected by significant depressive symptoms. The decreased health and limited cognitive ability of many nursing home residents makes treatment and research extremely challenging. This study will attempt to identify and implement treatments for depressed nursing home residents.

Participants are randomly assigned to receive either an active intervention or treatment as usual for 6 weeks. The active intervention is followed by 4 weeks of maintenance. The intervention is implemented primarily by existing nursing facility staff and focuses on increasing opportunities for residents to experience pleasant events through increased levels of activity and positive affect. The maintenance treatment involves incorporation of protocol-based activities into patient care plans. Patients have a follow-up visit 12 weeks after the study. Psychiatric evaluations, depression and mood rating scales, observed affect and activity participation, behavior problems, and staff burden are assessed.

ELIGIBILITY:
Inclusion Criteria:

* Nursing home residents
* DSM-IV criteria for major depressive disorder or dysthymia or Research Diagnostic Criteria for minor depressive disorder with current Geriatric Depression Scale scores > 11 and Mini Mental State scores >= 14

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2002-04; Primary Completion 2006-08 (Actual); Study Completion 2006-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Suzanne Meeks, PhD, Principal Investigator — University of Louisville
Locations (1):
- University of Louisville, Louisville, Kentucky, United States

IPD SHARING:
Plan to Share IPD: No